CLINICAL TRIAL: NCT02286700
Title: A Randomized, Double-Blind, Active Control, 5 Week Study to Evaluate the Safety and Skin Effects of A New, Twice-daily, Topically Applied Amino Acid Moisturizing Cream vs. Desonide Cream in Adult Atopic Dermatitis
Brief Title: Skin Effects of a Topical Amino Acid Moisturizing Cream and Desonide in Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeoStrata Company, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-ECD108
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Dermatitis, Atopic; Eczema
Keywords: dermatitis, eczema, itch, moisturizer, amino acid
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desonide Group (Active Comparator): Group randomly receiving desonide cream as the treatment cream for 3 weeks. Fifteen (15) gram tubes are dispensed at the beginning of each week and will be applied twice daily, by the subject, during the 3 week treatment phase.
  Interventions: Drug: Desonide Cream
- Amino Acid Group (Experimental): Group randomly receiving amino acid moisturizing cream as the treatment cream for 3 weeks. Fifteen (15) gram tubes are dispensed at the beginning of each week and will be applied twice daily, by the subject, during the 3 week treatment phase.
  Interventions: Other: Amino Acid Moisturizing Cream

INTERVENTIONS:
Drug: Desonide Cream — Study cream randomized and distributed to subjects, applied twice daily for 3 weeks and evaluated ability to reduce atopic dermatitis symptoms.
  Other Names: Desonide Cream 0.05%
  Arms: Desonide Group
Other: Amino Acid Moisturizing Cream — Study cream randomized and distributed to subjects, applied twice daily for 3 weeks and evaluated ability to reduce atopic dermatitis symptoms.
  Arms: Amino Acid Group

SUMMARY:
The purpose of this study is to compare the effects of an amino acid moisturizing cream and desonide cream in reducing skin symptoms associated with AD/eczema in subjects with mild to moderate atopic dermatitis/eczema.

DETAILED DESCRIPTION:
This is a double-blind, randomized study comparing the effects of an amino acid moisturizing cream and desonide cream in reducing skin symptoms associated with AD/eczema in subjects with mild to moderate atopic dermatitis/eczema. Atopic dermatitis (AD), also known as Eczema, is a chronic inflammatory skin disease that most commonly affects infants and children with a prevalence of 10-20% in children as compared to 1-3% in adults. Patients with AD have dry, irritated skin and often experience severe pruritus. Treatment of AD involves avoidance of triggers and infectious agents, cutaneous hydration, control of pruritus, and anti-inflammatory agents. Topical calcineurin inhibitors and steroids are commonly used prescription anti-inflammatory treatments. Unfortunately, there are potential side effects of long-term topical glucocorticoid use including skin atrophy, development of striae, perioral dermatitis, acne, and even hypothalamic-pituitary-adrenal axis suppression. However, many moisturizers are available without a prescription to soothe skin and reduce symptoms associated with AD/eczema via increased hydration, improved barrier function and anti-irritancy effects. The study cream being compared to desonide is a cosmetic moisturizing formulation that contains a cosmetic amino acid dipeptide (e.g., contains 2 amino acids). This study is being conducted to understand the benefits of the amino acid dipeptide moisturizing cream versus dermatologist-prescribed desonide cream in reducing the symptoms associated with AD/eczema in order to evaluate its potential use in the eczema care market. For this study, approximately 60 males and females, 18 years of age and older, who are in general good health, but diagnosed with mild to moderate AD/eczema, will be recruited, screened, and fully consented, with the goal of enrolling up to 42 evaluable subjects. The 42 Subjects (21 subjects per group) will be randomly and equally assigned to either one of 2 treatment groups of amino acid moisturizing cream or desonide cream. Neither study subjects nor study staff will be aware of the treatment assigned. The subjects will be asked to participate for approximately 5 weeks, over 5 study visits: Screening/Baseline, Weeks 1-3 (Treatment Period), Regression weeks 4 & 5. Each subject will receive one, 15 gram, blinded study cream at each treatment visit to apply twice daily at home for 3 weeks; a 2-week regression phase of no study cream will follow the treatment phase. A predetermined target lesion will be assessed at each time point via established clinical grading scales including: Target lesion Atopic Dermatitis Severity Index (TADSI), Eczema Area Severity Index (EASI), Static IGA of targeted lesion, Total IGA (PGA) and Body Surface Area involvement. All grading will be completed by the principal or sub-investigators. Photographs will also be taken at each time point to assess changes during the treatment and regression phases. Other established scales will be utilized to collect patient perception of skin effects such as: Patient-Oriented Eczema Measure (POEM), subjects' assessment of pruritus (VAS); a self-assessment questionnaire will be utilized to collect information on perceived benefits and product aesthetics. This study has been IRB approved and is scheduled to begin November of 2014 at Massachusetts General Hospital, specifically at the Clinical Unit for Research Trials in Skin (CURTIS) under principal investigator, Alexandra B. Kimball, MD. The study is being sponsored by NeoStrata Company, Inc, Princeton, NJ.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects in general good health 18 years of age or older
2. Diagnosis of atopic dermatitis will be made based on clinical criteria. Each patient must have at least one eczematous target lesion with area ranging from 10-500 cm2 of mild to moderate severity with a grade of at least 6 on the TADSI scale, plus presence of itch
3. Body surface area affected by AD lesions: ≤ 5% at start of treatment

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Any condition or therapy that in the investigator's opinion may pose a risk to the subject or that could interfere with any evaluation in the study
3. Widespread AD requiring systemic therapy
4. Diagnosis of allergic contact dermatitis
5. Known hypersensitivity to any of the constituents or excipients of the investigational product
6. Diagnosed with immunocompromised status
7. Use of systemic AD therapy, e.g. systemic corticosteroids, cyclosporine A, azathioprine, mycophenolate mofetil, or phototherapy in the past 1 month.
8. Use of phototherapy in the past 2 weeks
9. Use of any topical AD therapy such as corticosteroids or topical immunomodulators in the past 2 weeks
10. Use of local anti-itch or medical device treatments, e.g. benadryl, atopiclair, epiceram in the past 2 weeks
11. Use of topical moisturizers less than 24 hours in advance of the baseline visit on eczema lesions
12. Participation in another clinical research study with an investigational drug within 4 weeks before randomization in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in skin effects of an amino acid moisturizing cream and desonide cream in reducing skin symptoms associated with AD/eczema in subjects with mild to moderate atopic dermatitis/eczema. | 5 weeks
  Change in erythema, pruritus, exudation, excoriation and Lichenification from baseline of atopic dermatitis target lesions after application of either amino acid moisturizing cream or desonide cream twice daily for three weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kimball, MD, Principal Investigator — Massachusetts General Hospital: Clinical Unit for Research Trials in Skin
Locations (1):
- Mass General Hospital: Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

REFERENCES:
- [Background] Leung DM, Eichenfield LF, Boguniewicz M. Chapter 14. Atopic Dermatitis (Atopic Eczema). In: Goldsmith LA, Katz SI, Gilchrest BA, Paller AS, Leffell DJ, Wolff K. eds. Fitzpatrick's Dermatology in General Medicine, 8e. New York, NY: McGraw-Hill; 2012. http://accessmedicine.mhmedical.com/content.aspx?bookid=392&Sectionid=41138709. Accessed July 03, 2014.
- [Background] Elias PM, Steinhoff M. "Outside-to-inside" (and now back to "outside") pathogenic mechanisms in atopic dermatitis. J Invest Dermatol. 2008 May;128(5):1067-70. doi: 10.1038/jid.2008.88. PMID 18408746
- [Background] Williams HC. Clinical practice. Atopic dermatitis. N Engl J Med. 2005 Jun 2;352(22):2314-24. doi: 10.1056/NEJMcp042803. No abstract available. PMID 15930422
- [Background] Rudikoff D, Lebwohl M. Atopic dermatitis. Lancet. 1998 Jun 6;351(9117):1715-21. doi: 10.1016/S0140-6736(97)12082-7. No abstract available. PMID 9734903
- [Background] Langan SM, Williams HC. What causes worsening of eczema? A systematic review. Br J Dermatol. 2006 Sep;155(3):504-14. doi: 10.1111/j.1365-2133.2006.07381.x. PMID 16911274